CLINICAL TRIAL: NCT01028521
Title: Single-centre, Randomised, Double-blind, Placebo-controlled Clinical Study to Investigate Safety and Tolerability and Pharmacokinetics of Single Ascending Doses of CM3.1-AC100 in Healthy Male Volunteers
Brief Title: First in Man Clinical Study to Investigate Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of CM3.1-AC100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellMed AG, a subsidiary of BTG plc. (Industry)
Responsible Party: Dr. Peter Geigle, Cellmed AG
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: CellMed CM3.1-AC100/01; EudraCT No. 2009-017344-13 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-12-02; First posted 2009-12-09 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: First time in man, safety study, Cm3.1-AC100; Male volunteer aged 18 to 50 years at Screening

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM3.1-AC100 (Experimental)
  Interventions: Drug: CM3.1-AC100
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM3.1-AC100 — Solution for sc injection, single ascending doses
  Arms: CM3.1-AC100
Drug: Placebo — Solution for sc injection
  Arms: Placebo

SUMMARY:
A first time in man, phase I study to assess the safety, tolerability and pharmacokinetics of single ascending doses of CM3.1-AC100 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to any study specific procedures
* Body weight between 60.0 to 100.0 kg (both inclusive) and BMI 19 to 29.9 kg/m2 (both inclusive)
* Judged as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination)

Exclusion Criteria:

* Any history or presence of a clinically relevant disease as judged to be relevant by the Investigator
* Blood donation within 3 month before administration of the IP
* Have a history of hypersensitivity to the IP or any of the excipients or to medicinal products with similar chemical structures

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety measurements (Adverse events, ECG recordings, blood pressure, pulse, body temperature, laboratory variables,local tolerability, nausea questionnaire) | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Geigle, Dr. med., Study Chair — CellMed AG, a subsidiary of BTG plc.
Locations (1):
- Parexel International GmbH, Berlin, State of Berlin, Germany